CLINICAL TRIAL: NCT03743090
Title: Influence of Extracorporeal Circulation on the Development of OSA (Obstructive Sleep Apnea)
Status: Withdrawn | Type: Observational
Why Stopped: lack of PSG
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, FAHA, Head of Department, Astes
Other Study IDs: OSACS
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; obstructive sleep apnea
MeSH Terms: conditions — Coronary Artery Disease; Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CABG with ECC: Group of patients for whom CABG was performed under ECC. A polysomnography will be performed to all of these patients the day before surgery and the third postoperative day.
  Interventions: Diagnostic Test: Polysomnography.
- CABG without ECC: Group of patients for whom CABG was performed without ECC. A polysomnography will be performed to all of these patients the day before surgery and the third postoperative day.
  Interventions: Diagnostic Test: Polysomnography.

INTERVENTIONS:
Diagnostic Test: Polysomnography. — A polysomnography will be performed for all of the patients the day before surgery (value of reference), and on the second postoperative day (in order to examine the influence of ECC on the development of OSA).

SUMMARY:
* 1. Coronary artery bypass grafting (CABG) could be performed with or without extracorporeal circulation (ECC).
* 2. OSA (Obstructive Sleep Apnea) could be influenced by in intravenous perfusion.
* 3. ECC could influence the amount of intravenous perfusion administered to the patient.

The aim of this study was to examine the influence of ECC on the development of OSA.

DETAILED DESCRIPTION:
* 1. Coronary artery bypass grafting (CABG) could be performed with or without extracorporeal circulation (ECC).
* 2. OSA (Obstructive Sleep Apnea) could be influenced by in intravenous perfusion.
* 3. ECC could influence the amount of intravenous perfusion administered to the patient.

The aim of this study was to examine the influence of ECC on the development of OSA. The AHI (Apnea Hypopnea Index) will be used to assess this potential influence.

ELIGIBILITY:
Inclusion Criteria:

* All of the patients scheduled for an elective CABG

Exclusion Criteria:

* Patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All of the patients scheduled for an elective CABG at the Clinique Saint-Luc of Bouge (Namur, Belgium).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in the AHI | 3 days
  Change from baseline AHI (Apnea Hypopnea Index, which is the average amount of apnea and hypopnea per four of sleep) at the 3rd postoperative day. The AHI is derived from the polysomnography which will be performed to all of the patients the day before surgery and the 3rd postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Eric DEFLANDRE, MD, PhD, Principal Investigator — Astes

IPD SHARING:
Plan to Share IPD: No